CLINICAL TRIAL: NCT00796289
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled Study to Assess the Efficacy and Safety of Three Dosage Strengths of Pulsatile GnRH Delivered From a Iontophoretic Patch (Lutrepatch) Compared to Oral Treatment With Clomiphene Citrate or Placebo in Anovulatory or Oligoovulatory Infertile Females
Brief Title: Study to Assess the Efficacy and Safety of Three Dosage Strengths of Pulsatile GnRH Delivered From a Iontophoretic Patch Compared to Oral Treatment With Clomiphene or Placebo in Infertile Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-03
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
Keywords: anovulatory/oligoovulatory infertility
MeSH Terms: conditions — Infertility; Anovulation | interventions — Gonadotropin-Releasing Hormone; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- GnRH High Target Delivery (Experimental): 10 mg GnRH iontophoretic transdermal Lutrepatch with a high target delivery of pulsatile GnRH (every 90 minutes) for 21 days and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: GnRH iontophoretic transdermal Lutrepatch; Drug: placebo clomiphene citrate
- GnRH Medium Target Delivery (Experimental): 10 mg GnRH iontophoretic transdermal Lutrepatch with a medium target delivery of pulsatile GnRH (every 90 minutes) for 21 days and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: GnRH iontophoretic transdermal Lutrepatch; Drug: placebo clomiphene citrate
- GnRH Low Target Delivery (Experimental): 10 mg GnRH iontophoretic transdermal Lutrepatch with a low target delivery of pulsatile GnRH (every 90 minutes) for 21 days and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: GnRH iontophoretic transdermal Lutrepatch; Drug: placebo clomiphene citrate
- Clomiphene Citrate (Active Comparator): Placebo GnRH iontophoretic transdermal Lutrepatch with a high target delivery of pulsatile current (every 90 minutes) for 21 days and oral 50 mg clomiphene citrate for 5 days
  Interventions: Drug: clomiphene citrate; Drug: placebo GnRH patch
- Placebo (Placebo Comparator): Placebo GnRH iontophoretic transdermal Lutrepatch with a high target delivery of pulsatile current (every 90 minutes) for 21 days and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: placebo clomiphene citrate; Drug: placebo GnRH patch

INTERVENTIONS:
Drug: GnRH iontophoretic transdermal Lutrepatch — 10 mg GnRH iontopheretic transdermal patch. A new patch is applied two times each day (every 12 hours). Delivery current and membrane thickness adjusted to deliver the 'high target' study dose, which is estimated to be 800 picograms/ml
  Other Names: Lutrepatch; Gonadotropin-releasing hormone (GnRH)
  Arms: GnRH High Target Delivery
Drug: GnRH iontophoretic transdermal Lutrepatch — 10 mg GnRH iontopheretic transdermal patch. A new patch is applied two times each day(every 12 hours). Delivery current and membrane thickness adjusted to deliver the 'medium target' study dose, which is estimated to be 400-600 picograms/ml
  Other Names: Gonadotropin-releasing hormone (GnRH); Lutrepatch
  Arms: GnRH Medium Target Delivery
Drug: GnRH iontophoretic transdermal Lutrepatch — 10 mg GnRH iontopheretic transdermal patch. A new patch is applied two times each day (every 12 hours). Delivery current and membrane thickness adjusted to deliver the 'low target' study dose, which is estimated to be 200 picograms/ml
  Other Names: Gonadotropin-releasing hormone (GnRH); Lutrepatch
  Arms: GnRH Low Target Delivery
Drug: clomiphene citrate — Oral, 50 mg daily for 5 days
  Other Names: various tradenames
  Arms: Clomiphene Citrate
Drug: placebo clomiphene citrate — oral, taken for 5 days
  Arms: GnRH High Target Delivery; GnRH Low Target Delivery; GnRH Medium Target Delivery; Placebo
Drug: placebo GnRH patch — Placebo transdermal patch with a high target delivery of placebo(every 90 minutes). New patch to be applied every 12 hours.
  Arms: Clomiphene Citrate; Placebo

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of pulsatile GnRH delivered from a iontophoretic patch (Lutrepatch) for induction of ovulation in women with anovulatory/ oligoovulatory infertility, compared to placebo and to a reference treatment with clomiphene citrate.

ELIGIBILITY:
Inclusion Criteria:

1. Females between the ages of 18 and 38 years
2. Desire to become pregnant
3. Infertile due to ovulatory dysfunction as described below:

   * Unable to conceive for at least 1 year and
   * Anovulatory (defined as 4 or fewer menstrual cycles per year) or Oligo-ovulatory (defined as menstrual cycle frequency > 45 days)

Exclusion Criteria:

1. Requires donor oocytes or sperm
2. Two or more failed (defined as no biochemical pregnancy achieved) gonadotropin fertility treatment cycles - if previous gonadotropin success, no more than two failed subsequent cycles
3. Use of insulin-sensitizing drugs (e.g., Metformin) within 1 month prior to progesterone challenge

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | 30 days

SECONDARY OUTCOMES:
Pregnancy rate | 30 days
Incidence of Ovarian Hyperstimulation Syndrome (OHSS) | 30 days
Incidence of skin irritation | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (35):
- United States (35):
  - Watching Over Mothers and Babies Foundation, Tucson, Arizona
  - NEA Women's Clinic, Jonesboro, Arkansas
  - San Diego Fertility Center, San Diego, California
  - Compass Clinical Research, San Ramon, California
  - North Coast Women's Care Medical Group, Vista, California
  - Huntington Reproductive Center, Westlake Village, California
  - Florida Fertility Institute, Clearwater, Florida
  - All Women's Healthcare of Wesy Broward, Inc., Plantation, Florida
  - Atlanta Center for Reproductive Medicine, Atlanta, Georgia
  - Georgia Reproductive Specialists, Atlanta, Georgia
  - Women's Health Practice, Champaign, Illinois
  - University of Kentucky, Lexington, Kentucky
  - A Woman's Center for Reproductive Medicine, Baton Rouge, Louisiana
  - Maine Medical Center, Portland, Maine
  - Shady Grove Fertility Center, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hutzel Women's Health Specialists, Detroit, Michigan
  - CAREM Canadian American Reproductive Medicine, Hamtramck, Michigan
  - Women's Clinic of Lincoln, P.C., Lincoln, Nebraska
  - Fertility Center of Las Vegas, Las Vegas, Nevada
  - The Medical Group of Northern Nevada, Reno, Nevada
  - Women's Health Research Center LLC, Lawrenceville, New Jersey
  - Columbia University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Institute for Reproductive Health, Cincinnati, Ohio
  - Greater Cincinnati OB/GYN, Inc./Reproductive Medicine Research, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Clinical Trials of America Inc, Eugene, Oregon
  - Center for Health and Healing, Portland, Oregon
  - Greenville Hospital System, Greenville, South Carolina
  - Research Memphis Associates, LLC, Memphis, Tennessee
  - Center for Assisted Reproduction, Bedford, Texas
  - The Methodist Hospital, Houston, Texas
  - Center of Reproductive Medicine, Webster, Texas